CLINICAL TRIAL: NCT01768156
Title: Determination of the Prognostic and Predictive Value of the New Marker HE4 in Metastatic Ovarian Cancer Monitoring
Brief Title: Prognostic and Predictive Value of HE4 Biomarker in Metastatic Ovarian Cancer
Acronym: Meta-Four
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Meta-Four; 2010-A00152-37 (Registry Identifier: N° ID RCB)
Record Dates: First submitted 2013-01-09; First posted 2013-01-15 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Metastatic Ovarian Cancer
Keywords: ovarian cancer; biomarker; metastatic
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study arm (Experimental)
  Interventions: Other: Experimental arm

INTERVENTIONS:
Other: Experimental arm — Serum samples are collected:
  * at time of diagnosis of recurrence (before 1st chemotherapy)
  * during each cycle of chemotherapy
  * after the end of chemotherapy
  * every 3 month until treatment failure (3-6 samples)
  * stop at the progression or after 18 months post chemotherapy

SUMMARY:
HE4 is a new marker that could improve the detection of ovarian cancer. The HE4 assay may have an advantage over the CA-125 assay in that it is less frequently positive in patients with non malignant disease. Since the evaluation of HE4 for detection and diagnosis of ovarian cancer is well known, the behaviour of the marker during chemotherapy and follow-up period after treatment in metastatic ovarian cancer should be studied. It could be used in patient with non CA-125 secretary tumors. Prognosis and predictive value of HE4 should be compared with information provided by CA-125. The kinetics of HE4 values after treatment should be also analysed to determine the role that HE4 could play in the detection of recurrences during the follow-up of metastatic patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proved epithelial ovarian cancer (serous, mucinous, clear cell, endometrioid, undifferentiated type)
* Recurrence of anytime necessitating a new line of chemotherapy
* Patient having received adjuvant chemotherapy
* Informed consent signed prior any study specific procedures

Exclusion Criteria:

* More than 3 lines of chemotherapy
* Pregnancy or breastfeeding
* History of other cancers within the past 5 years (except curatively treated non-melanoma skin cancer and in situ cervical cancer)
* Psychological, social, geographical disorders or any other condition that would preclude study compliance (treatment modalities and study follow-up).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2010-09-24 (Actual); Primary Completion 2015-09-22 (Actual); Study Completion 2016-11-15 (Actual)

PRIMARY OUTCOMES:
To evaluate the predictive and prognostic value of HE4 marker | 18 months

SECONDARY OUTCOMES:
Determine the rate of patients without elevation of CA-125 presenting an elevation of HE4 that could be used for monitoring the disease. | 18 months

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut Bergonié, Bordeaux
  - CRLC Val d'Aurelle-Paul Lamarque, Montpellier